CLINICAL TRIAL: NCT06726187
Title: DSM-5 Personality Disorders in Adults with Autism
Status: Recruiting | Type: Observational
Sponsor: Parnassia Groep (Other)
Responsible Party: Sponsor
Other Study IDs: 2022.56
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Personality disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Personality Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 1: Adults with autism spectrum disorder
  Interventions: Other: Structured Clinical Interview for DSM-5 Screening Personality Questionnaire (SCID-5-SPQ).
- 2: The relative of the adult with autism spectrum disorder
  Interventions: Other: Structured Clinical Interview for DSM-5 Screening Personality Questionnaire (SCID-5-SPQ).

INTERVENTIONS:
Other: Structured Clinical Interview for DSM-5 Screening Personality Questionnaire (SCID-5-SPQ). — Screening questionnaire

SUMMARY:
Rationale: Self-report measures are frequently used for research and clinical assessments of adults with autism spectrum disorder (ASD). However, there has been little research examining agreement between self-report and informant-report in this population. Reliable self-report measures are essential for conducting research with and providing high quality clinical services for adults with autism spectrum disorder.

Objective: This study aims to examine the usefulness of self-report of DSM-5-TR PD traits in adults with ASD compared to informant-reports by administering the self-report screening measure of the Structured Clinical Interview for DSM-5 Screening Personality Questionnaire (SCID-5-SPQ).

ELIGIBILITY:
Inclusion criteria Inclusion criteria for ASD participants: (1) primary diagnosis of ASD according to the DSM-5-TR, (2) age 18+ years, (3) no intellectual disability, and (4) at least having completed a primary and secondary education.

Inclusion criteria for informants:

Participants were asked to identify individuals who knew them well and were capable of providing accurate descriptions of their personality traits, preferably informants that cohabited with the participants. When cohabitants were unavailable, participants were asked to identify "the person who knows you best." Additionally, eligibility of informants for inclusion required that, historically, the informant and the participant talked at least monthly and interacted face-to-face at least yearly.

Exclusion criteria Exclusion criteria for ASD participants: (1) no ASD diagnosis, (2) current substance abuse, (3) psychotic disorders, (4) schizophrenia, (5) eating disorder, (6), mental retardation (IQ<80), (7) suicidal ideations and (8) age <18 years.

Exclusion criteria for informants: (1) age <18 years, (2) intellectual disability, and (3) not being able to state and/or recognize psychological and problematic functioning of their participating relative with ASD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males and females (age ≥ 18 years), clinically diagnosed with ASD by a psychologist or a psychiatrist, without intellectual disability, and their informants. ASD participants will be recruited from Sarr Autism Rotterdam, the Netherlands, specialized in psychodiagnostic assessment and treatment for children, adolescents, and adults with ASD. Sarr is part of Parnassia Groep, multisite mental health institute in the Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Score SCID-5-PD | 1 day
  The main study parameters are the item scores on the SCID-5-PD.

CONTACTS AND LOCATIONS:
Locations (1):
- Sarr - Parnassia Groep Antes, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No